CLINICAL TRIAL: NCT05561062
Title: Combination of Atorvastatin and Mesalazine to Enhance Anti-inflammatory Effects and Attenuates Progression of Ulcerative Colitis
Brief Title: Atorvastatin in Patients With Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mostafa Bahaa, Teaching Assistant, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9/22021
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: double-blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): This group will take 1 g mesalamine three times daily
- Atorvastatin group (Active Comparator): This group will take 1 g mesalamine three times daily and atorvastatin 80 mg once daily
  Interventions: Drug: Atorvastatin 80mg

INTERVENTIONS:
Drug: Atorvastatin 80mg — Atorvastatin is one of the most effective drugs used to reduce intracellular cholesterol synthesis. it exerts numerous pleiotropic effects including anti-inflammatory, antioxidant properties, endothelial function improvement, and immunomodulation independent of its basic lipid-lowering properties
  Arms: Atorvastatin group

SUMMARY:
Ulcerative colitis (UC) is an idiopathic, chronic inflammatory disease characterized by diffused inflammation of the colon and rectum mucosa; however, the exact underlying mechanisms of UC remain poorly understood. Statins exert numerous pleiotropic effects including anti-inflammatory, antioxidant properties, endothelial function improvement, and immunomodulation independent of their basic lipid-lowering property.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Both male and female will be included
* Negative pregnancy test and effective contraception

Exclusion Criteria:

* Breastfeeding
* Significant liver and kidney function abnormalities
* Colorectal cancer patients
* Patients with severe UC
* Patients taking rectal or systemic steroids
* Patients taking immunosuppressives or biological therapies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Improvement in health related quality of life | 6 months
  HRQL questionnaire will be assessed according to a short-form (SF-36) questionnaire. The SF-36 is an indicator of overall health status and contains 10 items. The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100.

SECONDARY OUTCOMES:
changes in the level of inflammatory biomarkers | 6 months
  changes in the level of inflammatory biomarkers such as IL-6, fecal myeloperoxidase

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Mansoura University, Al Mansurah, Egypt

REFERENCES:
- [Derived] Alarfaj SJ, El-Haggar SM, Hegazy SK, Maher MM, Bahgat MM, Elmasry TA, Alrubia S, Alsegiani AS, Bahaa MM. Effect of a high dose atorvastatin as adjuvant therapy to mesalamine in attenuating inflammation and symptoms in patients with ulcerative colitis: a randomized controlled pilot study. Front Med (Lausanne). 2025 Jan 22;11:1490178. doi: 10.3389/fmed.2024.1490178. eCollection 2024. PMID 39911672